CLINICAL TRIAL: NCT05459155
Title: Effect of Synapse Medicine Decision Support on Inpatient Pharmacist Efficacy and Efficiency: a Hybrid Type 2 Implementation Study
Brief Title: Effect of Synapse Medicine Decision Support on Inpatient Pharmacist Efficacy and Efficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Synapse Medicine (Unknown); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Professor of Medicine, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P000659
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Infections; Heart Diseases; Lung Diseases; Kidney Diseases; Liver Diseases; Gastrointestinal Diseases
Keywords: Hospitalized Patients
MeSH Terms: conditions — Infections; Heart Diseases; Lung Diseases; Kidney Diseases; Liver Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective pre-post mixed methods hybrid type 2 effectiveness-implementation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist team post-intervention (Experimental): The direct subjects will be the inpatient pharmacists who round with general medicine teams and approve inpatient medication orders. They will be given full access to the Synapse Medicine medication decision support platform.
  Interventions: Other: Synapse medicine platform
- Pharmacist team pre-intervention (No Intervention): Pre-intervention, the inpatient pharmacists will round with general medicine teams and approve inpatient medication orders under conditions of usual care. They will base their recommendations on their knowledge and training and any tools (electronic or otherwise) that they choose to use.

INTERVENTIONS:
Other: Synapse medicine platform — Intervention is the Synapse medicine platform for inpatient pharmacists. This software analyzes drug-related risks based on each patient's clinical characteristics
  Arms: Pharmacist team post-intervention

SUMMARY:
Adverse drug events (ADE) are common and dangerous in the hospital and following discharge to the ambulatory setting. One cause of ADEs in both settings is medication regimen inappropriateness, including polypharmacy, drug-drug interactions, and medications that are inappropriate or inappropriately dosed given patients' age, renal, and hepatic function. Hospitalization provides a good opportunity to investigate medication appropriateness given new or worsening conditions and available expertise. Inpatient pharmacists are medication experts and often round with medical teams, but they may not always have all the information available at their fingertips to make optimal recommendations regarding medication appropriateness for each patient. Clinical decision support to pharmacists at the point of care has potential to improve the speed, quantity, and quality of medication recommendations to inpatient teams; any subsequent improvements to medication regimen appropriateness have the potential to reduce ADEs in the hospital and after discharge.

Specific Aims and Objectives

Aim 1: Implement real-time decision support regarding medication regimen appropriateness among pharmacists who round with inpatient medical teams.

Aim 2: Determine the effects of this intervention on the number of medication regimen recommendations and time spent per recommendation

Aim 3: Evaluate the use and usability of the decision support tool and develop strategies to mitigate barriers and promote facilitators of implementation using mixed methods implementation science approaches.

DETAILED DESCRIPTION:
This will be a prospective pre-post mixed methods hybrid type 2 effectiveness-implementation study. The study will take place at BWH and at Vanderbilt University Medical Center (VUMC). The direct subjects will be the inpatient pharmacists (4 at each site) who round with general medicine teams. Patients will be indirect subjects as pharmacists provide medication recommendations regarding these patients to the clinicians on each team with or without the Synapse software. We estimate this number of patients to be 3 new admitted patients per day per team x 56 days x 8 teams = 1344 patients (672 at MGB sites). Patients can be any patients admitted to these general medicine service teams at BWH and VUMC. The pharmacists are trained hospital pharmacists who round with general medicine service teams and approve inpatient medication orders. There are no local site restrictions. VUMC will cede IRB approval to the MGB IRB.

ELIGIBILITY:
Inclusion Criteria:

* any patient that the inpatient pharmacists care for on the inpatient medical team they round with

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in the number of medication recommendations made per patient | pre- and post-intervention periods: 4 weeks each per pharmacist
  Change from pre- to post-intervention in the number of recommendations regarding medication changes made by pharmacists per patient

SECONDARY OUTCOMES:
Change in the time spent per recommendation per patient | pre- and post-intervention periods: 4 weeks each per pharmacist
  Change from pre- to post-intervention in time spent per patient evaluating regimen appropriateness divided by the number of recommendations for that patient